CLINICAL TRIAL: NCT05015179
Title: Using Mixed Reality Technology to Facilitate Laparoscopic Partial Nephrectomy
Brief Title: Mixed Reality Technology in Laparoscopic Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Collaborators: Saint Petersburg State University, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 38/124-25
Record Dates: First submitted 2021-08-07; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Kidney Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Laparoscopic partial nephrectomy is performed with an intraoperative ultrasound (US) control
- Experimental (Experimental): Underwent Laparoscopic partial nephrectomy with the aid of the mixed reality model
  Interventions: Procedure: mixed reality technology in laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: mixed reality technology in laparoscopic partial nephrectomy — All patients undergo contrast-enhanced computed tomography before surgery. DICOM files are converted to a 3D model. This model is then sent to HoloLens 2 smart glasses using HLOIA software
  Arms: Experimental

SUMMARY:
The aim of our study was: a) to evaluate the usefulness of the MR model for renal pedicle exposure and identification of the tumor's exact location during LPN, and b) to evaluate the subjective utility of the MR model as an intraoperative reference tool.

Investigators prospectively enrolled 47 patients with LPN between June 2020 and February 2021. Patients were randomly assigned into two groups: the control group (24 patients), who underwent operation with an intraoperative ultrasound (US) control and the experimental group (23 patients), who underwent operation with the aid of the MR model. Randomization was performed using a computerized randomization program and sealed envelopes. Patients were included in the study if they were 18 years of age or older, were able to sign informed consent, and had T1a renal tumors amenable to LPN. Patients were excluded if they were unwilling to participate or did not meet the inclusion criteria. For each patient, investigators prospectively collected demographic data including age, body mass index, clinical tumor size, side, location, and complexity score according to the PADUA scoring system; perioperative data (including time for renal pedicle exposure and time for renal tumor detection and duration of ischemia); pathological data; data on postoperative functional outcome and complications, classified according to the Clavien-Dindo system.

ELIGIBILITY:
Inclusion Criteria:

* able to sign informed consent
* had T1a renal tumors amenable to LPN

Exclusion Criteria:

* were unwilling to participate
* did not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
time required to expose renal pedicle during laparoscopic partial nephrectomy | during operation completion, min
time required to get from renal pedicle to tumor during laparoscopic partial nephrectomy | during operation completion, min

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided